CLINICAL TRIAL: NCT03373994
Title: Tumor Perfusion and Hypoxia Evaluation and Comparation in 18F-FDG PET/CT
Brief Title: Perfusion and Hypoxia Evaluation in Tumors Using 18F-FDG PET/CT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Yingying Sun, Attending physician， doctor, Harbin Medical University
Other Study IDs: 14008
Record Dates: First submitted 2017-12-04; First posted 2017-12-14 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Perfusion and Hypoxia
Keywords: FDG, perfusion, hypoxia, tumor, PET
MeSH Terms: conditions — Hypoxia; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 18F-FDG PET/CT initial-time imaging: PET/CT imaging was underwent 5min after 18F-FDG injection.
  Interventions: Diagnostic Test: 18F-FDG PET/CT initial-time imaging
- 18F-FDG PET/CT balanced-time imaging: PET/CT imaging was underwent 60min after 18F-FDG injection.
  Interventions: Diagnostic Test: 18F-FDG PET/CT balanced-time imaging

INTERVENTIONS:
Diagnostic Test: 18F-FDG PET/CT initial-time imaging — 18F-FDG intravenous bolus injection after a fasting perid of more than 6 hours, simultaneously,PET/CT imaging using one bed lasting 5 minutes was underwent.
  Groups: 18F-FDG PET/CT initial-time imaging
Diagnostic Test: 18F-FDG PET/CT balanced-time imaging — 18F-FDG intravenous injection after a fasting perid of more than 6 hours. After 60 minutes, PET/CT imaging using 6-7 bed positions each lasting 2 minutes was underwent.
  Groups: 18F-FDG PET/CT balanced-time imaging

SUMMARY:
Investigators want to use 18F-FDG PET/CT imaging to reflect tumor perfusion and hypoxia.

DETAILED DESCRIPTION:
Perfusion and hypoxia were independent prognositic parameters for tumor patients. Developing a method that can evaluate tumor perfusion and hypoxia noninvasively and conveniently was in urgent need. 18F-FDG PET/CT imaging could reflect tumor hypoxia in 60min balanced imaging was proved and accepted. Moreover, FDG could diffuse out of the vasculature and through cell membranes passively and rapidly due to its lipophilicity, its regional uptake at initial times is expected to reflect tumor perfusion. So, investigators want to use 18F-FDG PET/CT imaging to evaluate tumor perfusion and hypoxia simutaniously，in order to guide the clinical diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1.solid tumor proved by pathology(d>3.0cm);
* 2.age>18-year-old;
* 3. Karnofsky performance status >70;
* 4.sign the informed consent.

Exclusion Criteria:

* 1.There are obvious metal implants near the tumor;
* 2.Can not lie still for 15 minutes.
* 3.Pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tumor patients aged more than 18 years with a histological confirmed diagnosis were eligible in our research. And all patients signed a written informed consent.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation of the distribution of FDG between initial-time and balanced-time PET/CT | 2018.1
  Initial-time and balanced-time PET/CT imaging were registrated using PET/CT Compare software in GE AW4.6 workstation. FDG distribution was evaluated in each imaging and the correlation was evaluated.

SECONDARY OUTCOMES:
SUVs in initial-time and balanced-time PET/CT | 2018.1
  the SUVmax and SUVmean was calculated in well-perfused area and hypoxia area in tumors using PET/CT Render software in GE AW4.6 workstation.

CONTACTS AND LOCATIONS:
Overall Officials: Baozhong Shen, Dr, Study Chair — The Fourth Hospital of Harbin Medical University
Locations (1):
- Yingying Sun, Harbin, Heil, China

IPD SHARING:
Plan to Share IPD: No